CLINICAL TRIAL: NCT04648007
Title: Diagnostic Ability of Plasma Based Neuromodulatory Cytokine Production (Kaihani Score) in Gambling Addiction
Brief Title: Validation of Kaihani Score for Gambling Addiction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Therapeutic Solutions International (Industry)
Responsible Party: Sponsor
Other Study IDs: TSOI-003
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Gambling Addiction
Keywords: addiction; BDNF
MeSH Terms: conditions — Gambling; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: 10 patients with no personal or family problems with gambling as assessed by the PG-YBOCS (obsessions-compulsions scale Yale-Brown (Y-BOCS), adapted for pathological gambling) (PG-YBOCS).
  Interventions: Diagnostic Test: Kaihani Score
- Moderate Gamblers: 10 patients with moderate gambling addiction as assessed by the PG-YBOCS (obsessions-compulsions scale Yale-Brown (Y-BOCS), adapted for pathological gambling) (PG-YBOCS).
  Interventions: Diagnostic Test: Kaihani Score
- Severe Gamblers: 10 patients with severe gambling addiction as assessed by the PG-YBOCS (obsessions-compulsions scale Yale-Brown (Y-BOCS), adapted for pathological gambling) (PG-YBOCS).
  Interventions: Diagnostic Test: Kaihani Score

INTERVENTIONS:
Diagnostic Test: Kaihani Score — Assessment of neuromodulatory chemicals in peripheral blood plasma samples.

SUMMARY:
The Kaihani Score is a blood based means of assessing molecules believed to be associated with gambling addiction.

The current clinical trial will assess the Kaihani Score in 3 groups:

Group 1: 10 patients with no personal or family problems with gambling as assessed by the PG-YBOCS (obsessions-compulsions scale Yale-Brown (Y-BOCS), adapted for pathological gambling) (PG-YBOCS).

Group 2: 10 patients with moderate gambling addiction as assessed by the PG-YBOCS (obsessions-compulsions scale Yale-Brown (Y-BOCS), adapted for pathological gambling) (PG-YBOCS).

Group 3: 10 patients with severe gambling addiction as assessed by the PG-YBOCS (obsessions-compulsions scale Yale-Brown (Y-BOCS), adapted for pathological gambling) (PG-YBOCS).

The goal of the study is to confirm preliminary efficacy of the Kaihani Score as a blood based means of assessing gambling propensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of pathological gambling (DSM IV criteria)
* First-time consultants.
* Without psychotropic treatment or treatment with a stable and unchanged for over a month.

Exclusion Criteria:

* Pregnant women and patients with hearing disorders
* Epilepsy (untreated or poorly balanced)
* Focal brain injury, whatever its origin (vascular, traumatic, tumor or infectious)
* History of head trauma with loss of consciousness,
* Administration of drugs or substances lowering the seizure threshold
* Sleep deprivation, jet lag, or drug withdrawal.
* Participants with a problem of uncorrected visual acuity.
* Other current addiction.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of 10 healthy volunteers, as well as 20 patients with gambling addictions. 10 of the patients will have moderate and 10 will have severe gambling addiction.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Kaihani Score | 1 Week
  Kaihani Score will be compared between non-gamblers, moderate gamblers, and severe gamblers.

CONTACTS AND LOCATIONS:
Overall Officials: James Veltmeyer, MD, Principal Investigator — Therapeutic Solutions International
Locations (1):
- Therapeutic Solutions International, Oceanside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided